CLINICAL TRIAL: NCT03943420
Title: One Research on Application of Key Technologies About Improving Cognitive Impairment Caused by Hypertension With the Therapy of Early Intervention With Qianyang Yuyin Granules
Brief Title: One Research on Improving Cognitive Impairment Caused by Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jiangsu Famous Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: BE2017770
Record Dates: First submitted 2019-01-29; First posted 2019-05-09 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-04

CONDITIONS: Hypertension
Keywords: Safety; Effectiveness; Therapy; Qianyang Yuyin Granules; Cognitive impairment; Hypertension
MeSH Terms: conditions — Hypertension; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Biospecimen Retention: Samples With DNA — Blood sample; Urine sample.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Experimental Group: Therapy A : Basic treatment + Qianyang Yuyin Granules
- Negative Control Group: Therapy B : Basic treatment
- Positive Control Group: Therapy C : Basic treatment + Donepezil

SUMMARY:
Using the therapy of early intervention with Qianyang Yuyin Granules to improve cognitive impairment caused by hypertension.

DETAILED DESCRIPTION:
Using the therapy of early intervention with Qianyang Yuyin Granules to improve cognitive impairment caused by hypertension.

The investigators designed a multi-center randomized controlled clinical trial to study the security and effectiveness of this therapy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 55 to 75 years old, male or female;
* Having a history of hypertension for more than 2 years but can maintain SBP ≤ 140 mmHg and BDP ≤ 90 mmHg with medication；
* 21 ≤ MMSE < 26, or 14 ≤ MoCA < 26, CDR < 0.5. Bseides, the chief complaint must happen after having hypertension；
* Meet TCM Syndrome Differentiation Standard：according to the Guidelines for the Clinical Research of Chinese Medicine New Drugs ( published by China Medical Science Press ) ：Overabundant liver-fire type：dizziness and headache, both face and eyes are red, dry mouth and bitter taste in mouth, red tongue with yellowish coating, wire and frequent pulse. Yin deficiency and yang hyperactivity type: dizziness and headache, Tinnitus and forgetfulness, sphoria with feverish sensation in chest & palms & soles, palpitation and insomnia, red tongue & thin white or less coating, wiry weak and numbered pulse；
* CTMRI hint: leukoaraiosis and no sign of Cerebral infarction；
* Patients or the guardian hold the right opinions over the research and are willing to obey researcher's orders；
* Having a certain degree of education (being able to read simple newspapers in the past)；
* Patients agree to sign informed consent。

Exclusion Criteria:

* Secondary hypertension；
* Taking certain kinds of antihypertensive drugs which may damage brain cognitive function；
* Diagnosed as depression or other mental disorders according to DSM-IV；
* Diagnosed as vascular dementia according to diagnostic criteria, CDR ≥ 0.5; alzheimer disease or dementia caused by some other reasons (including mixed dementia according to diagnostic criteria for VCI); cognitive impairment due to head injury。
* Suffering from certain kinds of diseases which may interfere the assessment of cognitive function, including those who are diagnosed as alcoholics and drugs or psychotropic medicine abusers during the last 5 years according to DSM-IV；
* Accompanied with severe neurological function disorder；
* Asthma, chronic severe primary cardiovascular disease, liver lesion, hematological lesions, lung diseases, diabetes or other severe diseases may influence the patients' survival such as cancer or AIDS；
* Other: Such as poor compliance, or can not attend the follow-up visit in time for some reasons；
* Taking the same kind of medicine during the last 30 days which may influence the trial；
* Is participating in another clinical study；
* Not up to TCM Syndrome Differentiation Standard。

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cognitive impairment caused by hypertension.
Sampling Method: Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2018-12-28 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Changes of brain image | 24 weeks
  Measure and record the volume changes of diseased alba, the micro-structure changes of alba fasciculus by MRI to see if the therapy effect or not.
Measure and assess the changes of VaDAS-cog ( Vascular Dementia Assessment Scale cognitive subscale ) among time points | 12 weeks, 24 weeks, 48 weeks
  Measure and record with VaDAS-cog

SECONDARY OUTCOMES:
Measure and assess the changes of MMSE ( Mini-mental State Examination ) among time points | 12 weeks, 24 weeks, 48 weeks
  Measure and record with MMSE
Measure and assess the changes of ADL ( Activity of Daily Living ) among time points | 12 weeks, 24 weeks, 48 weeks
  Measure and record with ADL
Measure and assess the changes of CDR ( Clinical Dementia Rating ) among time points | 12 weeks, 24 weeks, 48 weeks
  Measure and record with CDR
Incidence rate of outcome event | 24 weeks
  Record the outcome event and analyse the incidence rate
Therapeutic effect | 24 weeks
  Measure and record patients' systolic and diastolic blood pressure and analyse related data
Metabonomics | 24 weeks
  Measure and record the metabonomics ( Trx & TrxR ) index

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Province Hospital of Chinese Medcine, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided